CLINICAL TRIAL: NCT01817595
Title: Evaluation of Iphone Technology in Diabetes Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, Dr. Hugh Tildesley, Clinical Professor, Endocrine Research Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IBG star study
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Internet Blood Glucose Monitoring; iphone; meter
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG Star (Conventional Meter) (Active Comparator): 25 patients will use the (conventional) BG star meter in which patients will upload their readings onto a computer and send in their readings via email.
  Interventions: Other: BG Star Meter (Conventional) Internet Blood Glucose Reporting
- IBG Star Group (iPhone) (Active Comparator): 25 patients will be randomized to the iBGstar system will upload their readings to their iPhone and send in their readings using the iPhone.
  Interventions: Other: iBG Star (iphone) Internet Blood Glucose Method

INTERVENTIONS:
Other: BG Star Meter (Conventional) Internet Blood Glucose Reporting — Patients in BG Star Meter Group will report using BG software through uploading information onto a computer and sending readings to their endocrinologist via email
  Arms: BG Star (Conventional Meter)
Other: iBG Star (iphone) Internet Blood Glucose Method — 25 patients will be randomized to the iBGstar system will upload their readings to their iPhone and send in their readings using the iPhone.
  Arms: IBG Star Group (iPhone)

SUMMARY:
Background

With the emergence of the internet, health care professionals are changing the way they approach diabetes management. Internet Blood Glucose Monitoring Systems (IBGMS) are aimed at keeping blood glucose levels normal or in the range of acceptable levels to prevent the complications associated with diabetes. The Principal Investigators have completed a randomized clinical trial supporting the efficacy of IBGMS (1,2).

Patient satisfaction of reporting platform is essential to encourage patient reporting and participation in IBGMS. In this study, we wish to compare two different types of meters which will be used to internet blood glucose monitoring: the BG Star Meter (Conventional Meter), and the iBG Star Group (iPhone Technology).

Purpose and Rationale

Patients who are more satisfied with their meter and internet reporting platform are more likely to participate in an internet monitoring system. Patients often lack the motivation to report to their endocrinologist. With increased reporting to their healthcare professional, patients are more likely to benefit from such a system. This study aims to compare two types of meters and their respective internet reporting platforms to encourage patient participation.

Objectives

Our main goal is to compare the two types of meters.

Primary Outcomes Include:

1. Patient Satisfaction as measured by the "Diabetes Treatment Satisfaction Questionnaire" (DTSQ)
2. Frequency of reporting to endocrinologist
3. Number of Self-Monitoring Blood Glucose (SMBG) tests
4. Time taken to teach each patient the platforms

Research Design/Methods

Sample Size: 50 patients will be randomized into two groups:

BG Star Group (Conventional Meter) 25 patients will use the (conventional) BG star meter in which patients will upload their readings onto a computer and send in their readings via email.

IBG Star Group (iPhone Technology) 25 patients will be randomized to the iBGstar system will upload their readings to their iPhone and send in their readings using the iPhone.

Patients will be recruited from a Physician's private office.

Both the (Conventional meter) BG star and iBG star (iPhone Technology) group will be asked to perform SMBG 3 or more times per day and to upload their metered glucose values online every 2 weeks to be reviewed by the doctor.

Inclusion criteria:

* Type 1s
* Type 2s, can be on insulin, oral antihyperglycemic agents, or in combination.
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet Access

Exclusion criteria: Patients who do not meet the above criteria or are not willing to participate will not be included in the study.

DETAILED DESCRIPTION:
Background/Hypothesis

Management of diabetes is an evolving challenge to health care professionals. The fluctuations of glucose levels over the lifetime of patients with diabetes can lead to complications such as nephropathy, neuropathy, retinopathy and cardiovascular diseases. Although diabetes is a chronic disease, it can be controlled with use of medications (oral agents or insulin), and/or changes in life-style and diet.

With the emergence of the internet, health care professionals are changing the way they approach diabetes management. Internet Blood Glucose Monitoring Systems (IBGMS) are aimed at keeping blood glucose levels normal or in the range of acceptable levels to prevent the complications associated with diabetes. The Principal Investigators have completed a randomized clinical trial supporting the efficacy of IBGMS (1,2).

Patient satisfaction of reporting platform is essential to patient reporting and participation in IBGMS. In this study, we wish to compare two different types of meters which will be used to internet blood glucose monitoring: the BG Star Meter (Conventional Meter), and the iBG Star Group (iPhone Technology).

Purpose and Rationale

Patients who are more satisfied with their meter and internet reporting platform are more likely to participate in an internet monitoring system. Patients often lack the motivation to report to their endocrinologist. With increased reporting to their healthcare professional, patients are more likely to benefit from such a system. This study aims to compare two types of meters and their respective internet reporting platforms to encourage patient participation.

Objectives

Our main goal is to compare the two types of meters.

Primary Outcomes Include:

1. Patient Satisfaction as measured by the "Diabetes Treatment Satisfaction Questionnaire" (DTSQ)
2. Frequency of reporting to endocrinologist
3. Number of Self-Monitoring Blood Glucose (SMBG) tests
4. Time taken to teach each patient the platforms

Research Design/Methods

Sample Size: 50 patients will be randomized into two groups:

BG Star Group (Conventional Meter) 25 patients will use the (conventional) BG star meter in which patients will upload their readings onto a computer and send in their readings via email.

IBG Star Group (iPhone Technology) 25 patients will be randomized to the iBGstar system will upload their readings to their iPhone and send in their readings using the iPhone.

Patients will be recruited from a Physician's private office.

Both the (Conventional meter) BG star and iBG star (iPhone Technology) group will be asked to perform SMBG 3 or more times per day and to upload their metered glucose values online every 2 weeks to be reviewed by the doctor.

Inclusion criteria:

* Type 1s
* Type 2s, can be on insulin, oral antihyperglycemic agents, or in combination.
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet Access

Exclusion criteria: Patients who do not meet the above criteria or are not willing to participate will not be included in the study.

Confidentiality According to the guidelines of the University of British Columbia (UBC)/Providence Health Care Research Ethics Boards, the identity of participants will be kept confidential.

Data for each patient will be collected from the Clinical Research Coordinator and the Internet based glucose monitoring system. These data will only be accessed by the investigators and will be inputted into an Excel® spreadsheet where each patient will be given a unique identifier. All data pertaining to individual patients will be kept locked in the office of the study investigators.

Calculations and Statistics Statistical analysis will be performed on site by the researchers. Each group will complete the DTSQ. Questions revolve around satisfaction of treatment and are to be answered on a scale of 1 (very dissatisfied) to 6 (very Satisfied). Frequency of reporting will be determined through number of reports sent in per month. Total strip count will be recorded for each group. Time will be measured for the time it takes to train each patient in their respective meter/platform. All outcome measurements will be analysed using independent samples t-tests. Participants will only be identified by coded initials and a number to protect privacy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1s
* Type 2s, can be on insulin, oral antihyperglycemic agents, or in combination.
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet Access

Exclusion Criteria:

Patients who do not meet the above criteria or are not willing to participate will not be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 6 months
Frequency of SMBG testing | 6 months
Frequency of Reporting | 6 months
  How often patient sends report in to endocrinologist
Time required to teach meter/internet platform | Measured at beginning of study

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrine Research Society, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Tildesley HD, Mazanderani AB, Ross SA. Effect of Internet therapeutic intervention on A1C levels in patients with type 2 diabetes treated with insulin. Diabetes Care. 2010 Aug;33(8):1738-40. doi: 10.2337/dc09-2256. PMID 20668152
- See also: Related Info — http://www.diabetes.ca/documents/for-professionals/CJD--July_2011--H.Tildesley_.pdf